CLINICAL TRIAL: NCT04577963
Title: An Open-Label, Phase 1b/2 Study to Evaluate the Safety and Efficacy of Fruquintinib in Combination With Tislelizumab in Patients With Advanced Solid Tumors
Brief Title: A Study of Fruquintinib in Combination With Tislelizumab in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: At the time of study termination, both fruquintinib and tislelizumab are commercially available in the United States.
Sponsor: Hutchmed (Industry)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020-013-00US3
Record Dates: First submitted 2020-09-23; First posted 2020-10-08 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Triple Negative Breast Cancer; Endometrial Cancer; Solid Tumor, Unspecified, Adult; Colorectal Cancer
Keywords: Breast cancer; Triple negative; Her2-; HR-; ER-; PR-; Her2 negative; HR negative; ER negative; PR negative; TNBC; VEGF; VEGFR; Endometrial cancer; Colon; Rectal; mCRC; Colorectal
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Endometrial Neoplasms; Colorectal Neoplasms; Breast Neoplasms | interventions — HMPL-013; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): Approximately 6-12 patients with locally advanced or metastatic solid tumors will be enrolled to receive fruquintinib in combination with tislelizumab and assessed for DLTs during the 28-day DLT observation period
  Interventions: Drug: Fruquintinib; Drug: Tislelizumab
- Part 2 (Experimental): Patients will be enrolled to one of the following expansion cohorts:
  * Cohort A: TNBC (immuno-oncology [IO]-treated in the metastatic setting)
  * Cohort B: TNBC (IO-Naïve in the metastatic setting)
  * Cohort C: EC
  * Cohort D: MSS CRC
  Interventions: Drug: Fruquintinib; Drug: Tislelizumab

INTERVENTIONS:
Drug: Fruquintinib — Oral VEGFR inhibitor
  Other Names: HMPL-013
Drug: Tislelizumab — PD-1 inhibitor
  Other Names: BGB-A317

SUMMARY:
This is an open-label, multi-center, non-randomized, Phase 1b/2 study to assess the safety and efficacy of fruquintinib in combination with tislelizumab in patients with locally advanced or metastatic solid tumors. This study will be conducted in 2 parts; a Safety Lead-in Phase (Part 1) and a Dose Expansion Phase (Part 2).

The Safety Lead-in Phase, open to any-comer solid tumors, will determine the RP2D. The RP2D will be administered to 3 cohorts of patients in the Dose Expansion Phase.

* Cohort A: Advanced or Metastatic Triple Negative Breast Cancer (TNBC) (IO-treated)
* Cohort B: Advanced or Metastatic Triple Negative Breast Cancer (TNBC) (IO-Naïve)
* Cohort C: Advanced or Metastatic Endometrial Cancer (EC) (IO-Naïve)
* Cohort D: Advanced or Metastatic Colorectal Cancer (mCRC) (IO-Naïve)

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent signed by study patient or legally acceptable representative, as specified by health authorities and institutional guidelines;
2. Age ≥18 years;
3. Histologically or cytologically documented, advanced or metastatic Triple Negative Breast Cancer, histologically or cytologically documented, advanced or metastatic endometrial carcinoma, histologically or cytologically confirmed advanced or metastatic, unresectable adenocarcinoma of the colon or rectum.
4. Tumor tissue (archival or fresh tumor tissues as formalin-fixed paraffin-embedded blocks or approximately 15 unstained slides) for central laboratory assessment.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1.
6. At least 1 measurable lesion as defined by RECIST v1.1.

Exclusion Criteria:

1. Has at screening any central nervous system metastasis and/or leptomeningeal disease.
2. Except for Cohort A, Prior therapy targeting CTLA-4, PD-1, PD-L1 or programmed cell death protein ligand-2 (PD-L2) or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways.
3. Prior treatment with a VEGFR-TKI or anti-VEGFR antibody (eg, ramucirumab).
4. Except for Cohort D, prior treatment with an anti-VEGFR antibody (eg, bevacizumab).
5. Tumor tissue (archival or fresh tumor tissues as formalin-fixed paraffin-embedded blocks or approximately 15 unstained slides) for central laboratory assessment.
6. Active autoimmune diseases or history of autoimmune diseases that may relapse, or history of interstitial lung disease, noninfectious pneumonitis, or uncontrolled lung diseases including but not limited to pulmonary fibrosis, acute lung diseases, etc.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Schelman, MD, PhD, Study Director — HUTCHMED International
Locations (16):
- United States (16):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Highlands Oncology, Springdale, Arkansas
  - Beverly Hills Cancer Center, Beverly Hills, California
  - University of Colorado, Aurora, Colorado
  - Florida Cancer Specialists - FCS South, Port Charlotte, Florida
  - Florida Cancer Center North, St. Petersburg, Florida
  - Florida Cancer Specialists Panhandle, Tallahassee, Florida
  - Florida Cancer Specialists - East (FCS East), West Palm Beach, Florida
  - HOC AON Baton Rouge / Sarah Cannon, Baton Rouge, Louisiana
  - Messino Cancer Center, Asheville, North Carolina
  - Oklahoma University Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Tennessee Oncology-Chattanooga, Chattanooga, Tennessee
  - Tennesse Oncology, Nashville, Tennessee
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase 1b/2, 2-part, open-label study was conducted in patients with advanced or metastatic solid tumors.
Pre-assignment Details: The study consisted of a safety lead-in phase (Part 1) and a dose expansion phase (Part 2). A total of 52 patients were enrolled in this study (6 patients received study treatment in Part 1 and 46 patients received study treatment in Part 2). The study was terminated early based upon the strategic evaluation of clinical development of fruquintinib in the United States. This change was not based on any concern for patient safety or efficacy relative to fruquintinib and/or tislelizumab treatment.
Groups:
- Part 1: Solid Tumor of Any Type (IO-Treated/IO-Naïve in the Metastatic Setting): Patients with advanced or metastatic solid tumors of any type who had progressed on standard systemic therapy and for which no effective therapy or standard of care existed and who were either immuno-oncology (IO)-treated or IO-naïve in the metastatic setting were included in this cohort. Patients received fruquintinib 5 milligrams (mg) orally once daily (QD) for 3 weeks, followed by 1 week off in every 4-week cycle in combination with tislelizumab 300 mg intravenous (IV) infusion once every 4 weeks (Q4W) until radiologically determined progressive disease (PD) per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1, unacceptable toxicity, death, or withdrawal from study.
- Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting): Patients with advanced or metastatic triple negative breast cancer (TNBC) including those with estrogen receptor (ER) or progesterone receptor (PGR) low positive disease who had progressed on at least 1 line, but no more than 3 lines, of cytotoxic therapy in the locally advanced or metastatic setting and had progressed on prior immunotherapy in the metastatic setting were included in this cohort. Patients received fruquintinib 5 mg orally QD for 3 weeks, followed by 1 week off in every 4-week cycle in combination with tislelizumab 300 mg IV infusion Q4W until radiologically determined PD per RECIST v 1.1, unacceptable toxicity, death, or withdrawal from study.
- Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting): Patients with locally advanced or metastatic TNBC including those with ER or PGR low positive disease who had progressed on at least 1 line, but no more than 3 lines, of cytotoxic therapy in the locally advanced or metastatic setting and had not received prior therapy with an immune checkpoint inhibitor (ICI) or other immunotherapy in the metastatic setting were included in this cohort. Patients received fruquintinib 5 mg orally QD for 3 weeks, followed by 1 week off in every 4-week cycle in combination with tislelizumab 300 mg IV infusion Q4W until radiologically determined PD per RECIST v 1.1, unacceptable toxicity, death, or withdrawal from study.
- Part 2: Cohort C: EC (IO-Naïve): Patients with advanced or metastatic endometrial cancer (EC) who had progressed on 1 prior, platinum-based chemotherapy regimen for EC and had not received prior therapy with an ICI or other immunotherapy were included in this cohort. Patients received fruquintinib 5 mg orally QD for 3 weeks, followed by 1 week off in every 4-week cycle in combination with tislelizumab 300 mg IV infusion Q4W until radiologically determined PD per RECIST v 1.1, unacceptable toxicity, death, or withdrawal from study.
- Part 2: Cohort D: MSS mCRC (IO-Naïve): Patients with unresectable advanced or metastatic (m) microsatellite stable (MSS) colorectal cancer (CRC) who had failed 2 lines of standard chemotherapies, including fluorouracil, oxaliplatin, irinotecan and had received anti-vascular endothelial growth factor (VEGF) (if rat sarcoma [RAS]: wild-type tumor, mutated or status unknown) or endothelial growth factor receptor (EGFR) (if RAS wild-type tumor) antibody treatment were included in this cohort. Patients received fruquintinib 5 mg orally QD for 3 weeks, followed by 1 week off in every 4-week cycle in combination with tislelizumab 300 mg IV infusion Q4W until radiologically determined PD per RECIST v 1.1, unacceptable toxicity, death, or withdrawal from study.
Period: Part 1
Arm/Group | Part 1: Solid Tumor of Any Type (IO-Treated/IO-Naïve in the Metastatic Setting) | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) | Part 2: Cohort C: EC (IO-Naïve) | Part 2: Cohort D: MSS mCRC (IO-Naïve)
Started | 6 | 0 | 0 | 0 | 0
Completed (All patients from Part 1 were also included in the relevant Cohorts in Part 2 based on their tumor type [1 patient was included in Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) and 5 patients were included in Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting).) | 6 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1: Solid Tumor of Any Type (IO-Treated/IO-Naïve in the Metastatic Setting) | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) | Part 2: Cohort C: EC (IO-Naïve) | Part 2: Cohort D: MSS mCRC (IO-Naïve)
Started (Additional 46 unique patients were enrolled in Part 2 by tumor type.) | 0 | 1 (1 patient enrolled in Part 1 was also included in Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting).) | 11 (5 patients enrolled in Part 1 were also included in Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting).) | 1 | 39
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 11 | 1 | 39
Not completed — Death | 0 | 1 | 8 | 0 | 20
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 10
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 2
Not completed — Investigator decision | 0 | 0 | 0 | 0 | 1
Not completed — Sponsor terminated study | 0 | 0 | 3 | 1 | 4

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAS) included all enrolled patients who received at least 1 dose of fruquintinib or tislelizumab. 1 patient enrolled in Part 1 was also included in Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) and 5 patients enrolled in Part 1 were also included in Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting).
Groups:
- Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting): Patients with advanced or metastatic TNBC including those with ER or PGR low positive disease who had progressed on at least 1 line, but no more than 3 lines, of cytotoxic therapy in the locally advanced or metastatic setting and had progressed on prior immunotherapy in the metastatic setting were included in this cohort. Patients received fruquintinib 5 mg orally QD for 3 weeks, followed by 1 week off in every 4-week cycle in combination with tislelizumab 300 mg IV infusion Q4W until radiologically determined PD per RECIST v 1.1, unacceptable toxicity, death, or withdrawal from study.
- Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting): Patients with locally advanced or metastatic TNBC including those with ER or PGR low positive disease who had progressed on at least 1 line, but no more than 3 lines, of cytotoxic therapy in the locally advanced or metastatic setting and had not received prior therapy with an ICI or other immunotherapy in the metastatic setting were included in this cohort. Patients received fruquintinib 5 mg orally QD for 3 weeks, followed by 1 week off in every 4-week cycle in combination with tislelizumab 300 mg IV infusion Q4W until radiologically determined PD per RECIST v 1.1, unacceptable toxicity, death, or withdrawal from study.
- Part 2: Cohort C: EC (IO-Naïve): Patients with advanced or metastatic EC who had progressed on 1 prior, platinum-based chemotherapy regimen for EC and had not received prior therapy with an ICI or other immunotherapy were included in this cohort. Patients received fruquintinib 5 mg orally QD for 3 weeks, followed by 1 week off in every 4-week cycle in combination with tislelizumab 300 mg IV infusion Q4W until radiologically determined PD per RECIST v 1.1, unacceptable toxicity, death, or withdrawal from study.
- Part 2: Cohort D: MSS mCRC (IO-Naïve): Patients with unresectable advanced or metastatic MSS CRC who had failed 2 lines of standard chemotherapies, including fluorouracil, oxaliplatin, irinotecan and had received anti-VEGF (if RAS: wild-type tumor, mutated or status unknown) or EGFR (if RAS wild-type tumor) antibody treatment were included in this cohort. Patients received fruquintinib 5 mg orally QD for 3 weeks, followed by 1 week off in every 4-week cycle in combination with tislelizumab 300 mg IV infusion Q4W until radiologically determined PD per RECIST v 1.1, unacceptable toxicity, death, or withdrawal from study.
- Total: Total of all reporting groups
Arm/Group | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) | Part 2: Cohort C: EC (IO-Naïve) | Part 2: Cohort D: MSS mCRC (IO-Naïve) | Total
Number analyzed (Participants) | 1 | 11 | 1 | 39 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 8 | 0 | 32 | 40
  >=65 years | 1 | 3 | 1 | 7 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 11 | 1 | 12 | 25
  Male | 0 | 0 | 0 | 27 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 4 | 5
  Not Hispanic or Latino | 1 | 9 | 1 | 32 | 43
  Unknown or Not Reported | 0 | 1 | 0 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 2 | 3
  White | 1 | 10 | 1 | 31 | 43
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Patients With Dose-Limiting Toxicities (DLTs)
Description: According to National Cancer Institute Common Terminology Criteria for Adverse Events(AEs) v5.0, DLT was defined as any 1 of following toxicities during DLT assessment window and considered by Investigator to be related to 1 or more study treatments:a)Hematologic: grade(G) 4 neutropenia lasting >7 days, G ≥3 febrile neutropenia, G 3 thrombocytopenia with clinically significant bleeding, G 4 thrombocytopenia, G ≥4 anemia.b) Non-hematologic:all G ≥3 non-hematologic toxicities except:G 3 endocrinopathy controlled by hormonal replacement with no hospitalization and resolved to G ≤1 within 7 days, G 3 nausea/vomiting or diarrhea for <72 hours with antiemetic and supportive care, G 3 fatigue for <1 week, G ≥3 electrolyte abnormality lasting up to 72 hours and resolving with treatment, G 3 rash returning to baseline or G ≤1 within 7 days with treatment,G ≥3 amylase or lipase elevation without symptoms of pancreatitis,G 3 hypertension returning to baseline or G≤1 within 7 days with treatment.
Time Frame: From the first dose of study treatment (Day 1) up to Day 28 of Cycle 1 (cycle duration: 4 weeks)
Population: The DLT-evaluable analysis set included all patients enrolled in Part 1 of the study who received at least 1 dose of fruquintinib or tislelizumab and were considered DLT-evaluable based on the safety review committee review, according to the pre-specified criteria from the protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Solid Tumor of Any Type (IO-Treated/IO-Naïve in the Metastatic Setting): Patients with advanced or metastatic solid tumors of any type who had progressed on standard systemic therapy and for which no effective therapy or standard of care existed and who were either IO-treated or IO-naïve in the metastatic setting were included in this cohort. Patients received fruquintinib 5 mg orally QD for 3 weeks, followed by 1 week off in every 4-week cycle in combination with tislelizumab 300 mg IV infusion once Q4W until radiologically determined PD per RECIST v 1.1, unacceptable toxicity, death, or withdrawal from study.
Arm/Group | Part 1: Solid Tumor of Any Type (IO-Treated/IO-Naïve in the Metastatic Setting)
Number analyzed (Participants) | 6
Participants | 1

2. Primary Outcome: Part 1: Recommended Phase 2 Dose (RP2D) of Fruquintinib in Combination With Tislelizumab
Description: The RP2D of fruquintinib in combination with tislelizumab based on the safety and tolerability assessments in Part 1 patients.
Time Frame: From the first dose of study treatment (Day 1) up to Day 28 of Cycle 1 (cycle duration: 4 weeks)
Population: The SAS included all enrolled patients who received at least 1 dose of fruquintinib or tislelizumab. As pre-specified in SAP, all patients from Part 1 were also included in the relevant Cohorts in Part 2 based on their tumor type.
Measure: Number; unit: mg
Arm/Group | Part 1: Solid Tumor of Any Type (IO-Treated/IO-Naïve in the Metastatic Setting)
Number analyzed (Participants) | 6
mg | 5

3. Primary Outcome: Part 2: Objective Response Rate (ORR)
Description: The ORR was defined as the percentage of patients with a confirmed best overall response (BOR) of complete response (CR) or partial response (PR) as determined by the investigator using RECIST v1.1. The BOR was defined as the best response recorded from the start of study treatment until documented RECIST v1.1 progression or the start date of new anticancer therapy, whichever came first. The CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 millimeters (mm). The PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Tumor assessments performed every 8 weeks (+/-1 week) until PD, up to a maximum of approximately 34 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) | Part 2: Cohort C: EC (IO-Naïve) | Part 2: Cohort D: MSS mCRC (IO-Naïve)
Number analyzed (Participants) | 1 | 11 | 1 | 39
percentage of patients | 0 [NA to NA] — NA indicates that upper and lower limits of confidence interval (CI) were not estimable as there were no patients with CR or PR in that disease cohort. | 27.3 [6.0 to 61.0] | 0 [NA to NA] — NA indicates that upper and lower limits of confidence interval (CI) were not estimable as there were no patients with CR or PR in that disease cohort. | 5.1 [0.6 to 17.3]

4. Secondary Outcome: Part 1: Objective Response Rate
Description: The ORR was defined as the percentage of patients with a confirmed BOR of CR or PR as determined by the investigator using RECIST v1.1. The BOR was defined as the best response recorded from the start of study treatment until documented RECIST v1.1 progression or the start date of new anticancer therapy, whichever came first. The CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. The PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Tumor assessments performed every 8 weeks (+/-1 week) until PD, up to a maximum of approximately 34 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Part 1: Solid Tumor of Any Type (IO-Treated/IO-Naïve in the Metastatic Setting)
Number analyzed (Participants) | 6
percentage of patients | 16.7 [0.4 to 64.1]

5. Secondary Outcome: Parts 1 and 2: Progression-free Survival (PFS)
Description: PFS was defined as the time from the start of study treatment until the first radiographic documentation of objective progression as assessed by the investigator using RECIST v1.1, or death from any cause. The PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum also demonstrated an absolute increase of at least 5 mm. The appearance of 1 or more new lesions was also considered progression.
Time Frame: Tumor assessments performed every 8 weeks (+/-1 week) until PD, up to a maximum of approximately 34 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Solid Tumor of Any Type (IO-Treated/IO-Naïve in the Metastatic Setting) | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) | Part 2: Cohort C: EC (IO-Naïve) | Part 2: Cohort D: MSS mCRC (IO-Naïve)
Number analyzed (Participants) | 6 | 1 | 11 | 1 | 39
months | 3.8 [1.8 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | NA [NA to NA] — NA indicates that median, upper and lower limits of CI were not estimable due to insufficient number of patients with events at study closure. | 5.0 [1.8 to 7.4] | 5.5 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable for only 1 patient. | 3.6 [2.0 to 5.6]

6. Secondary Outcome: Parts 1 and 2: Disease Control Rate (DCR)
Description: The DCR was defined as the percentage of patients with a BOR of CR, PR, or stable disease (SD) lasting for at least 7 weeks as determined by the investigator using RECIST v1.1. The BOR was defined as the best response recorded from the start of study treatment until documented RECIST v1.1 progression or the start date of new anticancer therapy, whichever came first. The CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. The PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. The SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum on study.
Time Frame: Tumor assessments performed every 8 weeks (+/-1 week) until PD, up to a maximum of approximately 34 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Part 1: Solid Tumor of Any Type (IO-Treated/IO-Naïve in the Metastatic Setting) | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) | Part 2: Cohort C: EC (IO-Naïve) | Part 2: Cohort D: MSS mCRC (IO-Naïve)
Number analyzed (Participants) | 6 | 1 | 11 | 1 | 39
percentage of patients | 50.0 [11.8 to 88.2] | 0 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable due to no patients with CR, PR, or SD for at least 7 weeks. | 72.7 [39.0 to 94.0] | 100 [2.5 to 100] | 53.8 [37.2 to 69.9]

7. Secondary Outcome: Parts 1 and 2: Clinical Benefit Rate (CBR)
Description: The CBR was defined as the percentage of patients with a BOR of CR, PR, or durable SD (i.e., lasting for at least 6 months) as determined by the investigator using RECIST v1.1. Durable SD was SD for at least 6 months. The BOR was defined as the best response recorded from the start of study treatment until documented RECIST v1.1 progression or the start date of new anticancer therapy, whichever came first. The CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. The PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. The SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum on study.
Time Frame: Tumor assessments performed every 8 weeks (+/-1 week) until PD, up to a maximum of approximately 34 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Part 1: Solid Tumor of Any Type (IO-Treated/IO-Naïve in the Metastatic Setting) | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) | Part 2: Cohort C: EC (IO-Naïve) | Part 2: Cohort D: MSS mCRC (IO-Naïve)
Number analyzed (Participants) | 6 | 1 | 11 | 1 | 39
percentage of patients | 16.7 [0.4 to 64.1] | 0 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable due to no patients with CR, PR, or SD lasting for at least 6 months. | 27.3 [6.0 to 61.0] | 0 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable due to no patients with CR, PR, or SD lasting for at least 6 months. | 20.5 [9.3 to 36.5]

8. Secondary Outcome: Parts 1 and 2: Duration of Response (DoR)
Description: The DoR was defined as the time from the first occurrence of PR or CR by RECIST v1.1, whichever came first until PD or death. The CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. The PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. The PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum also demonstrated an absolute increase of at least 5 mm. The appearance of 1 or more new lesions was also considered progression.
Time Frame: Tumor assessments performed every 8 weeks (+/-1 week) until PD, up to a maximum of approximately 34 months
Population: The SAS included all enrolled patients who received at least 1 dose of fruquintinib or tislelizumab. As pre-specified in SAP, all patients from Part 1 were also included in the relevant Cohorts in Part 2 based on their tumor type. Only those patients with PR or CR (responders) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Solid Tumor of Any Type (IO-Treated/IO-Naïve in the Metastatic Setting) | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) | Part 2: Cohort C: EC (IO-Naïve) | Part 2: Cohort D: MSS mCRC (IO-Naïve)
Number analyzed (Participants) | 1 | 0 | 3 | 0 | 2
months | 14.9 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable for only 1 patient. |  | 14.9 [6.0 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. |  | NA [NA to NA] — NA indicates that median, upper and lower limits of CI were not estimable due to insufficient number of patients with events at study closure.

9. Secondary Outcome: Parts 1 and 2: Overall Survival (OS)
Description: The OS was defined as the time from start of study treatment until the date of death due to any cause.
Time Frame: From the first dose of study treatment (Day 1) up to date of death due to any cause, up to a maximum of approximately 34 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Solid Tumor of Any Type (IO-Treated/IO-Naïve in the Metastatic Setting) | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) | Part 2: Cohort C: EC (IO-Naïve) | Part 2: Cohort D: MSS mCRC (IO-Naïve)
Number analyzed (Participants) | 6 | 1 | 11 | 1 | 39
months | 16.4 [12.0 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | 25.8 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable for only 1 patient. | 14.1 [5.0 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | NA [NA to NA] — NA indicates that median, upper and lower limits of CI were not estimable due to insufficient number of patients with events at study closure. | 10.2 [7.1 to 11.7]

10. Secondary Outcome: Parts 1 and 2: Plasma Concentrations of Fruquintinib and Metabolite M11
Description: Blood samples were collected at the specified timepoints to determine plasma concentrations of fruquintinib and metabolite M11.
Time Frame: Pre-dose on Days 1, 8, 15, 21 of Cycle 1 and on Day 1 of Cycles 2, 4, 7, 13; 2 to 4 hours post-dose on Days 1 and 21 of Cycle 1 (cycle duration: 4 weeks)
Population: The pharmacokinetic (PK) analysis set included all patients with at least 1 quantifiable plasma or serum concentration of fruquintinib and/or tislelizumab. Only unique patients in Parts 1 and 2 were considered for PK analysis. Cohort A did not enroll any unique patients in Part 2. Only patients who had a quantifiable plasma/serum concentration of fruquintinib at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Part 1: Solid Tumor of Any Type (IO-Treated/IO-Naïve in the Metastatic Setting) | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) | Part 2: Cohort C: EC (IO-Naïve) | Part 2: Cohort D: MSS mCRC (IO-Naïve)
Number analyzed (Participants) | 1 | 0 | 6 | 1 | 37
nanograms per milliliter
  Fruquintinib: Cycle 1 Day 1: Pre-dose: number analyzed (Participants) | 1 | 0 | 6 | 1 | 36
  Fruquintinib: Cycle 1 Day 1: Pre-dose | 0 (0) |  | 0 (0) | 0 (0) | 0 (0)
  Fruquintinib: Cycle 1 Day 1: 2 to 4 hours post-dose | 5.49 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient. |  | 56.2 (52.9) | 125 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient. | 70.7 (34.3)
  Fruquintinib: Cycle 1 Day 8: Pre-dose: number analyzed (Participants) | 0 | 0 | 3 | 0 | 23
  Fruquintinib: Cycle 1 Day 8: Pre-dose |  |  | 222 (29.0) |  | 195 (57.0)
  Fruquintinib: Cycle 1 Day 15: Pre-dose: number analyzed (Participants) | 0 | 0 | 4 | 1 | 19
  Fruquintinib: Cycle 1 Day 15: Pre-dose |  |  | 240 (72.7) | 263 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient. | 177 (37.7)
  Fruquintinib: Cycle 1 Day 21: Pre-dose: number analyzed (Participants) | 1 | 0 | 3 | 0 | 16
  Fruquintinib: Cycle 1 Day 21: Pre-dose | 252 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient. |  | 216 (59.5) |  | 186 (51.4)
  Fruquintinib: Cycle 1 Day 21: 2 to 4 hours post-dose: number analyzed (Participants) | 1 | 0 | 1 | 0 | 10
  Fruquintinib: Cycle 1 Day 21: 2 to 4 hours post-dose | 327 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient. |  | 327 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient. |  | 267 (66.4)
  Fruquintinib: Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 0 | 0 | 3 | 1 | 18
  Fruquintinib: Cycle 2 Day 1: Pre-dose |  |  | 23.2 (15.3) | 15.2 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient. | 17.0 (17.7)
  Fruquintinib: Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 10
  Fruquintinib: Cycle 4 Day 1: Pre-dose |  |  | 5.12 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient. |  | 15.3 (8.89)
  Fruquintinib: Cycle 7 Day 1: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3
  Fruquintinib: Cycle 7 Day 1: Pre-dose |  |  |  |  | 28.6 (19.1)
  Fruquintinib: Cycle 13 Day 1: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Fruquintinib: Cycle 13 Day 1: Pre-dose |  |  |  |  | 12.3 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient.
  M11: Cycle 1 Day 1: Pre-dose: number analyzed (Participants) | 1 | 0 | 6 | 1 | 36
  M11: Cycle 1 Day 1: Pre-dose | 0 (0) |  | 0 (0) | 0 (0) | 0 (0)
  M11: Cycle 1 Day 1: 2 to 4 hours post-dose | 0 (0) |  | 0.415 (0.643) | 2.71 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient. | 0.413 (0.766)
  M11: Cycle 1 Day 8: Pre-dose: number analyzed (Participants) | 0 | 0 | 3 | 0 | 23
  M11: Cycle 1 Day 8: Pre-dose |  |  | 84.2 (53.5) |  | 60.7 (34.7)
  M11: Cycle 1 Day 15: Pre-dose: number analyzed (Participants) | 0 | 0 | 4 | 1 | 19
  M11: Cycle 1 Day 15: Pre-dose |  |  | 87.3 (32.4) | 139 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient. | 74.6 (45.9)
  M11: Cycle 1 Day 21: Pre-dose: number analyzed (Participants) | 1 | 0 | 3 | 0 | 16
  M11: Cycle 1 Day 21: Pre-dose | 148 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient. |  | 106 (40.0) |  | 66.1 (28.0)
  M11: Cycle 1 Day 21: 2 to 4 hours post-dose: number analyzed (Participants) | 1 | 0 | 1 | 0 | 10
  M11: Cycle 1 Day 21: 2 to 4 hours post-dose | 124 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient. |  | 124 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient. |  | 69.1 (25.4)
  M11: Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 0 | 0 | 3 | 1 | 18
  M11: Cycle 2 Day 1: Pre-dose |  |  | 30.8 (12.6) | 40.5 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient. | 20.5 (14.4)
  M11: Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 10
  M11: Cycle 4 Day 1: Pre-dose |  |  | 16.6 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient. |  | 19.3 (10.4)
  M11: Cycle 7 Day 1: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3
  M11: Cycle 7 Day 1: Pre-dose |  |  |  |  | 31.4 (8.60)
  M11: Cycle 13 Day 1: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  M11: Cycle 13 Day 1: Pre-dose |  |  |  |  | 11.7 (NA) — NA indicates that standard deviation (SD) was not estimable for 1 patient.

11. Secondary Outcome: Parts 1 and 2: Serum Concentrations of Tislelizumab
Description: Blood samples were collected at the specified timepoints to determine serum concentrations of tislelizumab.
Time Frame: Pre-infusion on Day 1 of Cycles 1, 2, 4, 7, 13; at end of infusion on Day 1 of Cycles 1 and 4; on Days 8, 15, and 21 of Cycle 1 (cycle duration: 4 weeks)
Population: The PK analysis set included all patients with at least 1 quantifiable plasma or serum concentration of fruquintinib and/or tislelizumab. Only unique patients in Parts 1 and 2 were considered for PK analysis. Cohort A did not enroll any unique patients in Part 2. Only patients who had a quantifiable plasma/serum concentration of tislelizumab at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Part 1: Solid Tumor of Any Type (IO-Treated/IO-Naïve in the Metastatic Setting) | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) | Part 2: Cohort C: EC (IO-Naïve) | Part 2: Cohort D: MSS mCRC (IO-Naïve)
Number analyzed (Participants) | 6 | 0 | 6 | 1 | 37
micrograms per milliliter
  Cycle 1 Day 1: Pre-infusion | 0 (0) |  | 0 (0) | 0 (0) | 0 (0)
  Cycle 1 Day 1: End of infusion: number analyzed (Participants) | 5 | 0 | 6 | 1 | 36
  Cycle 1 Day 1: End of infusion | 105 (23.5) |  | 101 (22.7) | 74.0 (NA) — NA indicates that SD was not estimable for 1 patient. | 78.3 (19.9)
  Cycle 1 Day 8: number analyzed (Participants) | 5 | 0 | 4 | 1 | 34
  Cycle 1 Day 8 | 49.5 (12.7) |  | 54.4 (15.1) | 45.2 (NA) — NA indicates that SD was not estimable for 1 patient. | 39.2 (10.0)
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 0 | 4 | 1 | 32
  Cycle 1 Day 15 | 34.3 (11.2) |  | 31.4 (7.63) | 36.7 (NA) — NA indicates that SD was not estimable for 1 patient. | 27.7 (8.72)
  Cycle 1 Day 21: number analyzed (Participants) | 3 | 0 | 4 | 0 | 26
  Cycle 1 Day 21 | 27.3 (13.1) |  | 28.1 (6.58) |  | 20.3 (5.58)
  Cycle 2 Day 1: Pre-infusion: number analyzed (Participants) | 5 | 0 | 4 | 1 | 30
  Cycle 2 Day 1: Pre-infusion | 22.2 (8.27) |  | 19.3 (10.5) | 21.5 (NA) — NA indicates that SD was not estimable for 1 patient. | 15.1 (5.14)
  Cycle 4 Day 1: Pre-infusion: number analyzed (Participants) | 3 | 0 | 3 | 1 | 21
  Cycle 4 Day 1: Pre-infusion | 29.9 (11.8) |  | 41.0 (15.5) | 46.6 (NA) — NA indicates that SD was not estimable for 1 patient. | 25.1 (8.64)
  Cycle 4 Day 1: End of infusion: number analyzed (Participants) | 3 | 0 | 2 | 1 | 20
  Cycle 4 Day 1: End of infusion | 158 (47.6) |  | 172 (7.78) | 137 (NA) — NA indicates that SD was not estimable for 1 patient. | 114 (25.4)
  Cycle 7 Day 1: Pre-infusion: number analyzed (Participants) | 1 | 0 | 2 | 0 | 8
  Cycle 7 Day 1: Pre-infusion | 57.2 (NA) — NA indicates that SD was not estimable for 1 patient. |  | 50.0 (31.0) |  | 35.5 (14.4)
  Cycle 13 Day 1: Pre-infusion: number analyzed (Participants) | 1 | 0 | 1 | 0 | 3
  Cycle 13 Day 1: Pre-infusion | 45.9 (NA) — NA indicates that SD was not estimable for 1 patient. |  | 26.0 (NA) — NA indicates that SD was not estimable for 1 patient. |  | 34.9 (7.32)

12. Secondary Outcome: Parts 1 and 2: Number of Patients With Antidrug Antibodies (ADAs) to Tislelizumab
Description: Blood samples were collected at the specified timepoints to detect ADAs to tislelizumab. Treatment-induced ADA was defined as ADA negative at baseline and ADA positive post-baseline. Treatment-boosted ADA was defined as ADA positive at baseline that was boosted to a 4-fold or higher-level following treatment administration.
Time Frame: From the first dose of study treatment (Day 1) up to end of treatment, up to approximately 17 months for Part 1 and 20 months for Part 2
Population: The ADA analysis set included all patients who received at least 1 dose of tislelizumab and had a baseline and at least 1 post-baseline ADA result. As pre-specified in SAP, all patients from Part 1 were also included in the relevant Cohorts in Part 2 based on their tumor type.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Solid Tumor of Any Type (IO-Treated/IO-Naïve in the Metastatic Setting) | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) | Part 2: Cohort C: EC (IO-Naïve) | Part 2: Cohort D: MSS mCRC (IO-Naïve)
Number analyzed (Participants) | 6 | 1 | 10 | 1 | 29
Participants
  Treatment-Induced ADA | 2 | 0 | 3 | 0 | 10
  Treatment-Boosted ADA | 0 | 0 | 0 | 0 | 2

13. Secondary Outcome: Part 2: Number of Patients With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs) and TEAEs Leading to Treatment Discontinuation
Description: An AE was any untoward medical occurrence in a clinical study patient temporally associated with the use of a study treatment, whether or not considered related to the treatment. An AE was considered "serious" if, in the view of either the investigator or sponsor, it resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, was a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, was an abnormal pregnancy outcome in a child born to a female patient/female partner of a male patient exposed to study treatment or was an important medical event. TEAEs were AEs that started or worsened in severity on or after the first dose of study treatment and up to 30 days after the date of last study treatment administration.
Time Frame: From the first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment, approximately 21 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) | Part 2: Cohort C: EC (IO-Naïve) | Part 2: Cohort D: MSS mCRC (IO-Naïve)
Number analyzed (Participants) | 1 | 11 | 1 | 39
Participants
  TEAEs | 1 | 11 | 1 | 39
  TESAEs | 0 | 2 | 1 | 20
  TEAEs leading to fruquintinib treatment discontinuation | 1 | 1 | 1 | 9
  TEAEs leading to tislelizumab treatment discontinuation | 1 | 1 | 0 | 9

14. Secondary Outcome: Part 2: Change From Baseline in Programmed Death-Ligand 1 (PD-L1) Expression
Description: Expression of PD-L1 biomarker was planned to be assessed in tumor tissues of the patients. Baseline was defined as the last non-missing assessment prior to the first administration of any study treatment (whichever occurred first), including scheduled and unscheduled visits, unless otherwise specified.
Time Frame: Baseline (Day 1) up to end of treatment, up to approximately 20 months
Population: The SAS included all enrolled patients who received at least 1 dose of fruquintinib or tislelizumab. Based upon the strategic evaluation of clinical development of fruquintinib in the United States, the study was early terminated prior to data collection for this outcome measure.
Arm/Group | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) | Part 2: Cohort C: EC (IO-Naïve) | Part 2: Cohort D: MSS mCRC (IO-Naïve)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment, approximately 18 months for Part 1 and 21 months for Part 2. All-cause mortality (deaths) were collected from Day 1 up to end of follow up, approximately 34 months.
Description: The SAS included all enrolled patients who received at least 1 dose of fruquintinib or tislelizumab. As pre-specified in SAP, all patients from Part 1 were also included in the relevant Cohorts in Part 2 based on their tumor type. Therefore, the results presented by Cohort for Part 2 are inclusive of Part 1.
Arm/Group | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) | Part 2: Cohort C: EC (IO-Naïve) | Part 2: Cohort D: MSS mCRC (IO-Naïve)
All-Cause Mortality (participants affected / at risk) | 1/1 | 8/11 | 0/1 | 20/39
Serious Adverse Events (participants affected / at risk) | 0/1 | 2/11 | 1/1 | 20/39
Other Adverse Events (participants affected / at risk) | 1/1 | 11/11 | 1/1 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) (N=1) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) (N=11) | Part 2: Cohort C: EC (IO-Naïve) (N=1) | Part 2: Cohort D: MSS mCRC (IO-Naïve) (N=39)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Malignant ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 1 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 2
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 2: Cohort A: TNBC (IO-Treated in the Metastatic Setting) (N=1) | Part 2: Cohort B: TNBC (IO-Naïve in the Metastatic Setting) (N=11) | Part 2: Cohort C: EC (IO-Naïve) (N=1) | Part 2: Cohort D: MSS mCRC (IO-Naïve) (N=39)
Diarrhoea (Gastrointestinal disorders) | 0 | 6 | 0 | 10
Nausea (Gastrointestinal disorders) | 0 | 4 | 0 | 9
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 7
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 7
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 7
Constipation (Gastrointestinal disorders) | 0 | 3 | 0 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oral discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 5 | 1 | 26
Oedema peripheral (General disorders) | 0 | 2 | 0 | 2
Influenza like illness (General disorders) | 0 | 0 | 0 | 3
Chills (General disorders) | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 9
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 9
Weight decreased (Investigations) | 0 | 3 | 0 | 5
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 6
Amylase increased (Investigations) | 0 | 1 | 0 | 6
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 0 | 5
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0 | 6
Lipase increased (Investigations) | 0 | 2 | 0 | 5
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 4
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 3
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 2 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 3
Platelet count decreased (Investigations) | 1 | 1 | 0 | 1
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 0 | 2
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 2
Thyroxine free increased (Investigations) | 0 | 2 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 2
Blood calcium increased (Investigations) | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 1 | 0 | 0
Low density lipoprotein increased (Investigations) | 0 | 1 | 0 | 0
Protein total increased (Investigations) | 0 | 1 | 0 | 0
Thyroxine increased (Investigations) | 0 | 1 | 0 | 0
Tri-iodothyronine free increased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 0 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 4 | 1 | 13
Hypotension (Vascular disorders) | 0 | 0 | 0 | 3
Jugular vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 3 | 0 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 3
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 3 | 0 | 11
Hypothyroidism (Endocrine disorders) | 0 | 3 | 0 | 11
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 5
COVID-19 (Infections and infestations) | 0 | 2 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 3
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 6
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 5
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early based upon the strategic evaluation of clinical development of fruquintinib in the United States. This change was not based on any concern for patient safety or efficacy relative to fruquintinib and/or tislelizumab treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT04577963/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT04577963/SAP_001.pdf